CLINICAL TRIAL: NCT06707025
Title: The Expression of CD24 "do-not-eat-me" Signal in Cholangiocarcinoma
Acronym: CD24CCA
Status: Active, not recruiting | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Eithan Galun, Principal Investigator, Hadassah Medical Organization
Other Study IDs: 0520-23-HMO; Israel ministry of health (Other: Israel ministry of health)
Record Dates: First submitted 2024-11-10; First posted 2024-11-27 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-10

CONDITIONS: Cholangiocarcinoma
Keywords: CD24; Human; Liver cancer; MiR122
MeSH Terms: conditions — Cholangiocarcinoma; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — the investigators are collecting plasma circulating free DNA. the investigators are not performing DNA sequencing. this is similar to chipSEQ.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The investigators found an inverse relationship between CD24 and MiR-122 levels. Then the investigators found that CD24 that goes up with MiR-122 down makes macrophages unable to engulf the tumor cells. All this in mice. the investigators are interested in confirming this result in humans. Details of the preliminary results are attached to the submission of the research documents. the investigators will compare Cholangiocarcinoma tumors with other solid tumors, including liver tissue. The need to deepen understanding the investigators will also make a comparison between cancerous tissue and "normal" tissue adjacent to the tumor.

DETAILED DESCRIPTION:
The investigators will collect samples from the tissue bank. All materials will be kept in refrigerators at minus 80, except for the sections of the paraffin blocks at room temperature. The source of some of the biological samples and the information accompanying them in this study is Midgem - the Israeli repository for biological samples for research. Midgem is a non-profit association that operates within the Ministry of Health as an infrastructure for the promotion of bioresearch - Medical and industrial in Israel. The donors to Midgem are patients with malignant diseases, Non-malignant diseases as well as healthy volunteers. In Midgem, residues are collected from tissues already removed during surgery/taking a biopsy and/or samples from blood/saliva/urine/other body fluids donations and the accompanying medical information required for use in legally approved studies.There is no risk to the donors as a result of the donation of the samples and information and their use, since the donation is transferred to Midgem only after it has been ascertained beyond any doubt that the ability of the diagnosis and/or treatment of the donors will not be harmed. All the information transferred to the researchers is coded, in such a way that the investigators do not allow the identification of the donors' details. Since the donors to Midgem have signed a consent form for the collection and storage of samples and information for use in any legally approved study, the investigators request an exemption from signing a dedicated informed consent form for this study. The samples and information transferred to this study are donated in accordance with what is detailed in the inclusion criteria for the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Donors with cholangiocarcinoma samples

Exclusion Criteria:

* Donors who do not have cholangiocarcinoma samples

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver cancer.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2026-10-28 (Estimated)

PRIMARY OUTCOMES:
the investigators will analyze ductular reaction and cancer stem cells markers including CD24, CD44 | All along the study, from the first recruitment to the last recruitment. average of 1 year
  the investigators will perform the analysis on tissue samples of cholangiocarcinoma and non tumor controls, using immunohistochemistry and RT-PCR

CONTACTS AND LOCATIONS:
Overall Officials: Tamar Hamburger, Study Chair — Hadassah Hospital Hebrew University
Locations (1):
- Hdassah Hospital, Jerusalem, Israel, Israel

IPD SHARING:
Plan to Share IPD: Yes
Publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: January 2028 for 7 years
Access Criteria: After publication any one.
URL: https://www.eithangalun.com/